CLINICAL TRIAL: NCT00005704
Title: Pharmacologic Intervention for Postcessation Weight Gain
Status: Completed | Type: Observational
Sponsor: University of Memphis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4359; R18HL045057 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To test pharmacologic intervention for smoking postcessation weight gain using nicotine gum and phenylpropanolamine (PPA).

DETAILED DESCRIPTION:
BACKGROUND:

Despite the potential importance of weight gain to smoking relapse, in 1991 there had been virtually no success in eliminating, or even reducing, the weight gain following smoking cessation. Two promising pharmacologic methods for reducing postcessation weight gain were nicotine gum and an over-the-counter drug, phenylpropanolamine gum ([PPA]. However, the relative efficacy of these two drugs had never been evaluated and the mechanisms of action of both drugs on weight gain were unknown.

DESIGN NARRATIVE:

The investigators determined the efficacy of nicotine gum and phenylpropanolamine (PPA) gum relative to a placebo in the reduction of postcessation weight gain throughout a 13-week combined behavioral and pharmacologic treatment program. Following cessation of the drugs at the end of treatment, they monitored long-term effects of these drugs on body weight at both a 6- and a 12-month follow-up. They also determined the mechanism of action of both nicotine gum and PPA gum (viz., changes in dietary intake, physical activity, or metabolic rate) on change in weight during the course of treatment and evaluated withdrawal symptoms of smoking cessation as they were moderated by either nicotine gum or PPA gum use during the course of treatment. Finally, they investigated whether PPA and nicotine gum produced an incremental effect on smoking cessation (relative to placebo gum) in a sample of female smokers who were at high risk for postcessation weight gain at posttest and at a 6- and 12-month follow-up.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-07; Study Completion 1997-06

REFERENCES:
- [Background] Klesges RC, Mealer CZ, Klesges LM. Effects of alcohol intake on resting energy expenditure in young women social drinkers. Am J Clin Nutr. 1994 Apr;59(4):805-9. doi: 10.1093/ajcn/59.4.805. PMID 8147323
- [Background] Klesges RC, Ray JW, Klesges LM. Caffeinated coffee and tea intake and its relationship to cigarette smoking: an analysis of the Second National Health and Nutrition Examination Survey (NHANES II). J Subst Abuse. 1994;6(4):407-18. doi: 10.1016/s0899-3289(94)90334-4. PMID 7780298
- [Background] Klesges RC, Klesges LM. The relationship between body mass and cigarette smoking using a biochemical index of smoking exposure. Int J Obes Relat Metab Disord. 1993 Oct;17(10):585-91. PMID 8242127
- [Background] Camp DE, Klesges RC, Relyea G. The relationship between body weight concerns and adolescent smoking. Health Psychol. 1993 Jan;12(1):24-32. doi: 10.1037//0278-6133.12.1.24. PMID 8462495
- [Background] Klesges RC, Shelton ML, Klesges LM. Effects of television on metabolic rate: potential implications for childhood obesity. Pediatrics. 1993 Feb;91(2):281-6. PMID 8424001
- [Background] Rushing PA, Winders SE, Watson SL, Klesges RC. Acute administration of phenylpropanolamine fails to affect resting energy expenditure in men of normal weight. Obes Res. 1997 Sep;5(5):470-3. doi: 10.1002/j.1550-8528.1997.tb00673.x. PMID 9385624
- [Background] Meyers AW, Klesges RC, Winders SE, Ward KD, Peterson BA, Eck LH. Are weight concerns predictive of smoking cessation? A prospective analysis. J Consult Clin Psychol. 1997 Jun;65(3):448-52. doi: 10.1037//0022-006x.65.3.448. PMID 9170768
- [Background] Klesges RC, Winders SE, Meyers AW, Eck LH, Ward KD, Hultquist CM, Ray JW, Shadish WR. How much weight gain occurs following smoking cessation? A comparison of weight gain using both continuous and point prevalence abstinence. J Consult Clin Psychol. 1997 Apr;65(2):286-91. doi: 10.1037//0022-006x.65.2.286. PMID 9086692
- [Background] Eck LH, Bennett AG, Egan BM, Ray JW, Mitchell CO, Smith MA, Klesges RC. Differences in macronutrient selections in users and nonusers of an oral contraceptive. Am J Clin Nutr. 1997 Feb;65(2):419-24. doi: 10.1093/ajcn/65.2.419. PMID 9022525
- [Background] Klesges RC, Eck LH, Ray JW. Who underreports dietary intake in a dietary recall? Evidence from the Second National Health and Nutrition Examination Survey. J Consult Clin Psychol. 1995 Jun;63(3):438-44. doi: 10.1037//0022-006x.63.3.438. PMID 7608356
- [Background] Klesges RC, Debon M, Ray JW. Are self-reports of smoking rate biased? Evidence from the Second National Health and Nutrition Examination Survey. J Clin Epidemiol. 1995 Oct;48(10):1225-33. doi: 10.1016/0895-4356(95)00020-5. PMID 7561984
- [Background] Klesges RC, Klesges LM, DeBon M, Shelton ML, Isbell TR, Klem ML. Effects of phenylpropanolamine on withdrawal symptoms. Psychopharmacology (Berl). 1995 May;119(1):85-91. doi: 10.1007/BF02246058. PMID 7675954
- [Background] Hultquist CM, Meyers AW, Whelan JP, Klesges RC, Peacher-Ryan H, DeBon MW. The effect of smoking and light activity on metabolism in men. Health Psychol. 1995 Mar;14(2):124-31. doi: 10.1037//0278-6133.14.2.124. PMID 7789347
- [Background] Audrain JE, Klesges RC, Klesges LM. Relationship between obesity and the metabolic effects of smoking in women. Health Psychol. 1995 Mar;14(2):116-23. doi: 10.1037//0278-6133.14.2.116. PMID 7789346